CLINICAL TRIAL: NCT01681394
Title: Effect of the Administration of a Polyphenol-rich Cocoa Extract on Peripheral Blood Mononuclear Cells Gene Expression in Humans
Brief Title: Effect of a Polyphenol-rich Cocoa Extract on Peripheral Blood Mononuclear Cells Gene Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PBMCS-CTNS-01
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Cardiovascular Function; Gene Expression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Product 1 (Active Comparator): 250 g of chocolate cream supplemented with 2.3 g of polyphenol-rich cocoa extract (containing 1050 mg of total polyphenols)
  Interventions: Dietary Supplement: Polyphenol-rich cocoa extract
- Control product (Placebo Comparator): 250 g of chocolate cream
  Interventions: Dietary Supplement: Chocolate cream

INTERVENTIONS:
Dietary Supplement: Polyphenol-rich cocoa extract — 250 g of chocolate cream supplemented with 2.3 g of polyphenol-rich cocoa extract (containing 1050 mg of total polyphenols)
  Arms: Product 1
Dietary Supplement: Chocolate cream
  Arms: Control product

SUMMARY:
It has been evidenced that chocolate and cocoa consumption increase vasodilation and reduce blood pressure. However, the mechanisms implicated in these effects have not been elucidated yet. The purpose of this study is to evaluate changes in gene expression induced by the administration of a polyphenol-rich cocoa extract in peripheral blood mononuclear cells (PBMC) in humans.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, double-blind and cross-over study. The intervention will consist in the administration of 250g of chocolate cream with or without the extract after 12 hours fasting. Blood samples will be taken at point 0, 2, 3 and 6 hours after the administration. At each time point, blood pressure and endothelial function (with a non-invasive method) will be measured.

ELIGIBILITY:
Inclusion Criteria:

1.Healthy males between the ages of 20 and 39 who do not meet any of the exclusion criteria.

Exclusion Criteria:

1. Body mass index (BMI) lower than 18 or greater than 27 Kg/m2
2. Smokers
3. Regular medication
4. Consumption of medication during the last week
5. Following a weight-loss diet
6. Vegetarians
7. Abnormal glucose levels
8. Diabetes
9. Cardiovascular disease
10. Gastrointestinal disease
11. Anemia
12. Allergy

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Gene expression changes in PBMCs (using a microarray) | 0-6 hours

SECONDARY OUTCOMES:
Blood pressure | 0-2-3-6 hours
Endothelial function (assessed by ischemic reactive hyperemia) | 0-2-3-6 hours
Plasma levels of procyanidins metabolites | 0-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, PhD, Principal Investigator — University Rovira i Virgili
Locations (1):
- Technological Center of Nutrition and Health (CTNS), Reus, Tarragona, Spain